CLINICAL TRIAL: NCT02732223
Title: Complementary Therapy of Omega 3 Fatty Acids, Plant Sterols and Polyphenols Over Cardiovascular Markers in Statin Treated Patients
Brief Title: Combined Bioactive Therapy Effects Over Cardiovascular Markers in Statin Treated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Adriana Bertolami, MD. PhD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: NºCAAE 27349114.5.3001.0067
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases
Keywords: Atherosclerosis; omega 3; plant sterols; polyphenols
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional treatment (Experimental): Daily functional treatment consisted of seven fish oil softgels (1.7g EPA+DHA), two dark chocolate truffles containing plant sterol esters and two green tea sachets.
  Interventions: Dietary Supplement: Functional treatment
- Control treatment (Placebo Comparator): Control treatment consisted of seven soy bean oil softgels, two regular dark chocolate truffles and two anise tea sachets
  Interventions: Dietary Supplement: Control treatment

INTERVENTIONS:
Dietary Supplement: Functional treatment — Omega 3 fatty acids, plant sterols and polyphenols
  Arms: Functional treatment
Dietary Supplement: Control treatment — placebo supplements
  Arms: Control treatment

SUMMARY:
Atherosclerosis, one major cause of morbidity and mortality worldwide, is a complex and multifactorial disease triggered especially due to high level of plasma lipids and that involves three mainly conditions: chronic inflammation, dyslipidemia and oxidative stress. Taking into account the high costs of disease management, eminent suboptimal response and low compliance to drug therapies, the combined use of natural bioactive compound able to reduce atherosclerosis risk could provide an additional protection. In this study, the effects of three bioactive components, namely omega-3 fatty acids, plants sterols and polyphenols present in green tea, will be evaluated over atherosclerosis biomarkers in individuals with dyslipidemia controlled by drugs. It will be carried out a randomized, double-blind, placebo-controlled, crossover clinical study, with participation of 70 subjects. At each intervention period, study participants will receive a packaged for the functional or placebo treatment. Functional treatment packaged will be composed by omega 3 softgels (fish oil), a chocolate containing plant sterols and green tea. Placebo treatment will be composed by corn oil softgels, regular chocolate, and anise tea. Subjects will be advised to consume the softgels and chocolate twice a day after main meals and to drink two cups of tea per day. After evaluation of inflammation, dyslipidemia and oxidative stress biomarkers, subjects with the greatest response to the functional treatment will be selected for additional 6 weeks of functional intervention associated to a reduction of the hypolipidaemic drugs intake, which will be prescribed individually after evaluation of the responsible physician.

DETAILED DESCRIPTION:
From eligible subjects, 70 participants will be recruited for a first visit, when they will give informed consent. Also at the first visit, medical reports will be confirmed by each participant, anthropometric measures will be recorded and blood samples will be collected. After first blood analysis results, participants with stable parameters will be called for a second visit when they will be enrolled in a randomized, placebo-controlled, crossover trial, with 4 treatment periods of 6 weeks each, corresponding to a total of 7 visits. At each visit, blood samples and anthropometric measures will be collected. At the first intervention period, study participants will receive a packaged for the functional or control treatment. Functional treatment packaged will be composed by omega 3 softgels (fish oil), chocolate containing plant sterols and green tea. Control treatment will be composed by soy oil softgels, regular chocolate, and anise tea. Subjects will be advised to consume 3 softgels and 1 chocolate twice a day, after main meals, and to drink two cups of tea per day. After a 6-weeks washout period (third visit), the groups will be switched (crossover) and participants will receive the functional or control treatment for more 6 weeks (fourth visit). After biomarkers evaluation, the subjects with the greatest response to the functional treatment will be selected for additional 6 weeks of functional intervention associated to a reduction of the hypolipidaemic drugs (statin) dosage, which will be prescribed individually and by the evaluation of the responsible physician.

ELIGIBILITY:
Inclusion Criteria:

* The primary selection criteria were current statin (simvastatin or atorvastatin) and hypoglycemic treatment (metformin and/or gliclazide).

Exclusion Criteria:

* Exclusion criteria were patients who were taking omega 3 fatty acids, plant sterol or green tea supplements; uncontrolled diabetes (HbA1c > 7.5%) or dyslipidemia (LDL-C > 100 mg/dL); pregnant females; and patients who presented any congenital cardiac disorders, uncontrolled endocrine, renal or hepatic disease and excessive alcohol consumption.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
LDL | after 6 weeks of supplementation
C-reactive protein | after 6 weeks of supplementation
Malondialdehyde | after 6 weeks of supplementation

SECONDARY OUTCOMES:
Omega 3 fatty acids profile | after 6 weeks of supplementation
  plasma samples
Cholesterol synthesis and absorption markers | after 6 weeks of supplementation
  plasma samples
Antioxidant enzymes activity | after 6 weeks of supplementation
  Lysates samples

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Scolaro B, Nogueira MS, Paiva A, Bertolami A, Barroso LP, Vaisar T, Heffron SP, Fisher EA, Castro IA. Statin dose reduction with complementary diet therapy: A pilot study of personalized medicine. Mol Metab. 2018 May;11:137-144. doi: 10.1016/j.molmet.2018.02.005. Epub 2018 Feb 20. PMID 29503145